CLINICAL TRIAL: NCT01328769
Title: Febuxostat, Blood Pressure and the Intrarenal Renin-Angiotensin System (RAS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paul N. Hopkins (Other)
Responsible Party: Sponsor-Investigator, Paul N. Hopkins, Professor of Internal Medicine, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 42916
Record Dates: First submitted 2011-03-29; First posted 2011-04-05 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
Keywords: uric acid; febuxostat; hypertension; intra-renal renin-angiotensin system; renal plasma flow; angiotensin II
MeSH Terms: conditions — Hypertension | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat (Active Comparator): Investigational
  Interventions: Drug: Febuxostat
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat
  Arms: Febuxostat
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this study the investigators will recruit hypertensive subjects with higher than average uric acid levels to test the effect of lowering uric acid with febuxostat on several measures as listed below. This will be a randomized, double-blind, placebo-controlled, parallel group study.

DETAILED DESCRIPTION:
Persons with hypertension (HTN) often have higher uric acid than normotensives, especially in hypertensives with metabolic syndrome.1-5 Recent prospective studies also suggest that persons with higher uric acid are at greater risk to develop hypertension.4-7 Uric acid in childhood appears to be particularly predictive of both early-onset hypertension and blood pressure later in life.4, 5, 8 While many had considered elevated uric acid as merely a marker for increased renal sodium reabsorption, recent data suggests a potentially causal role. Rats made mildly hyperuricemic by treatment with the uricase inhibitor oxonic acid become hypertensive. The increase in blood pressure in these rats was blocked by administration of renin-angiotensin system (RAS) blockers or by reduction of uric acid with allopurinol.9 More recently, febuxostat was also shown effective in this experimental model.10 Febuxostat was recently approved by the FDA as Uloric. Febuxostat is a xanthine oxidase (XO) inhibitor (like the older drug allopurinol), and is indicated for the chronic management of hyperuricemia in patients with gout.

The investigators have reported a clear relationship between higher serum uric acid and increased intrarenal angiotensin II as assessed by intravenous angiotensin II (Ang II) infusions in human subjects.11 In this model, the change in renal blood flow in response to infused Ang II serves as an indirect indicator of renal vascular exposure to endogenous Ang II. In the setting of high endogenous intrarenal Ang II, renovascular AT1 receptors are down-regulated and the normal reduction in renal blood flow in response to infused exogenous Ang II becomes blunted. The investigators found that increased serum uric acid is strongly correlated to blunting of the normal response to infused Ang II. Other studies by our colleagues in Boston have demonstrated that treatment with ACE inhibitors or angiotensin receptor blockers restores normal responsiveness to infused Ang II in hypertensives with this blunted response and that such patients may be particularly responsive to RAS blockade.12-14 The studies in rats and our results with the association of uric acid suggest that elevated uric acid may cause an increase in intrarenal Ang II or otherwise interact with Ang II and thereby promote hypertension. In this study, the investigators propose to explore the causality of uric acid in affecting blood pressure and, importantly, to begin to explore the underlying mechanism of such a response using our unique protocol in human subjects.

Recent results from a randomized cross-over study of 30 hyperuricemic, hypertensive adolescents showed that allopurinol (200 mg twice daily) resulted in a significant reduction in blood pressure as compared with placebo.4, 15, 16 However, similar studies in adults are lacking and no study has provided insights into mechanisms whereby uric acid might raise blood pressure in humans. Endothelial dysfunction was consistently improved by allopurinol treatment in patients with congestive heart failure17, 18 and several other conditions.19 It would be of great scientific and clinical interest if a mechanistic role for uric acid in adult hypertension could be demonstrated. The investigators have a unique opportunity to examine uric acid as a contributor to overactivity of the intrarenal RAS and impaired nitric oxide production. The investigators hypothesize that hypertensives with elevated uric acid will experience a significant fall in uric acid in response to administration of febuxostat which will correlate with an improvement in vascular responses to infused Ang II, and improved endothelial function.

As part of the same protocol the investigators will be able to assess the effect of febuxostat on proximal and distal sodium clearance by using uric acid clearance as a surrogate for proximal tubular sodium absorption. Uric acid reabsorption is indirectly coupled to sodium reabsorption: anions enter proximal tubular cells via a sodium-coupled electroneutral system and anions are then exchanged for urate.20 Renal uric acid clearance is directly and closely correlated with renal lithium clearance, a well-validated measure of proximal tubular sodium reabsorption, and both clearances have been used to estimate proximal tubular sodium handling in large, population-based studies,21, 22 as well as to measure acute responses to, for example, insulin infusion,23 beta-blocker treatment,24 and volume expansion.20, 25 Other studies have found decreased proximal tubular uric acid or lithium clearance associated with a positive family history of hypertension26 and with an adducin gene variant associated with hypertension.27 In summary, the investigators will examine the effects of lowering uric acid with febuxostat on both intrarenal RAS activity as measured by renovascular response to Ang II infusion, and on proximal tubular sodium absorption as measured by uric acid clearance. Potential effects on endothelial function, arterial stiffness, and blood pressure will also be tested.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hypertension. For purposes of this study, the investigators define mild to moderate hypertension as being on no more than 1-2 antihypertensive medications and blood pressure <140 mm Hg systolic and <90 mm Hg diastolic based on mean seated blood pressure at the screening visit in our clinic. For these visits, the investigators measure blood pressure using a Dinamap automatic oscillometric cuff while subjects are seated quietly. The subjects are left in a quiet room without speaking for 5 minutes initially. The Dinamap is started and the technician leaves the room and 3 blood pressures are obtained at intervals of 2 minutes. The investigators use the mean of last 2 blood pressures for classification purposes. This is the approach the investigators have used in several multicenter studies including HyperGEN and the NHLBI Family Heart Study.
* Age 18 to 60.
* Uric acid =5.8 mg/dl. This was the mean uric acid among hypertensives in our prior study.11 As renal plasma flow response to Ang II infusion decreased linearly with higher uric acid, the investigators felt that using higher than average uric acid will provide greater power.

Exclusion Criteria:

* Severe or poorly controlled hypertension (treated blood pressure >160 mm Hg systolic or >100 mm Hg diastolic).
* Diabetes (type 1 or type 2).
* Estimated GFR <60 ml/min.
* Persons unable stop all medications (including antihypertensives) other than stable doses of thyroxine or estrogen for at least 2 weeks.
* Secondary hypertension.
* Prior history of clinically diagnosed coronary artery disease or congestive heart failure.
* Taking uric acid lowering medication within 1 month of screening visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul N Hopkins, Principal Investigator — Cardiovascular Genetics
Locations (1):
- Cardiovascular Genetics, University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Febuxostat: 80mg once daily
- Placebo: Matching placebo dose 80mg once daily
Period: Overall Study
Arm/Group | Febuxostat | Placebo
Started | 25 | 24
Completed | 25 | 23
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Febuxostat: 80mg daily
- Total: Total of all reporting groups
Arm/Group | Febuxostat | Placebo | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (8.1) | 48.6 (8.0) | 49.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Renal Plasma Flow in Response to Infused Angiotensin II
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Error); unit: ml/minute
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 25 | 23
ml/minute | -54.1 (13.4) | -10.8 (14)

2. Secondary Outcome: Change in Endothelial Function
Description: Endothelial function was calculated by software from the manufacturer VENDYS. The measurement was taken by using the index of area under the curve of the finger temperature recovery curve just after releasing a blood pressure cuff. The blood pressure cuff occluded blood flow for 5 minutes as compared to the temperature curve in the non-occluded arm.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: ratio of finger temperature
Arm/Group | Febuxostat | Placebo
Number analyzed (Participants) | 18 | 18
ratio of finger temperature | 1.66 (0.63) | 1.90 (0.39)

ADVERSE EVENTS:
Arm/Group | Febuxostat | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No